CLINICAL TRIAL: NCT00060333
Title: Phase II Trial Evaluating Resection Followed By Adjuvant Radiation Therapy (RT) For Patients With Desmoplastic Melanoma
Brief Title: Adjuvant Radiation Therapy in Treating Patients With Resected Desmoplastic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0275; NCI-2009-00641 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000301633 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-01

CONDITIONS: Recurrent Melanoma
Keywords: recurrent melanoma; stage I melanoma; stage II melanoma; stage III melanoma
MeSH Terms: conditions — Melanoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (adjuvant radiation therapy) (Experimental): Within 8 weeks after surgical resection, patients undergo radiation therapy twice weekly over approximately 2.5 weeks for a total of 5 fractions in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
This phase II trial is studying how well adjuvant radiation therapy works in treating patients who have undergone surgery for desmoplastic melanoma. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving radiation therapy after surgery may kill any tumor cells remaining after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the recurrence rates in patients with desmoplastic melanoma (DM) >= 1 mm deep treated with adjuvant radiotherapy after surgical resection.

II. Assess recurrence rates in patients with locally recurrent DM treated with adjuvant radiotherapy after surgical resection.

SECONDARY OBJECTIVES:

I. Evaluate the impact of adjuvant radiation therapy after surgical resection on disease free and overall survival.

II. Evaluate the immediate and long-term morbidity of the addition of radiotherapy to surgery.

OUTLINE:

Within 8 weeks after surgical resection, patients undergo radiation therapy twice weekly over approximately 2.5 weeks for a total of 5 fractions in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria

* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Pathologically proven DM >= 1 mm in depth or locally recurrent DM; recurrent tumor is defined as a tumor found =< 2 cm from the previous excision or within the surgical bed (which includes the extent of previous skin flaps)
* DM resected with pathologically negative margins; acceptable surgery includes standard wide local excision and Moh's surgery

  * Tumors on the trunk proximal extremities need to have a >= 2 cm negative margin; tumors located on the head and neck and distal extremities will have an attempt at 2 cm negative margins but due to location and subsequent concern regarding cosmesis a margin < 2 cm will be acceptable if margin is negative
  * Margins from tumors resected using the Moh's technique will be accepted if negative and best approximation of tumor width will be made
* Radiation therapy (RT) is to begin =< 8 weeks after definitive surgical resection
* Adjuvant systemic therapy (immunotherapy or chemotherapy) must be postponed until irradiation is completed

Exclusion Criteria

* Previous irradiation to the same site
* Non-healing surgical wound
* Active infection at the surgical site
* Evidence of metastatic disease; local nodal disease is still eligible for the trial
* Life expectancy < 1 year
* Melanoma with focally desmoplastic features, in which the desmoplastic melanoma is not the predominant histologic pattern of the tumor, will be excluded; non-desmoplastic neurotropic melanoma and non-desmoplastic spindle cell melanoma are also excluded
* Previous malignancy < 5 years excluding basal cell carcinoma or squamous cell carcinoma of the skin or cervical carcinoma in situ (with the exception of patients who have stage I breast cancer who were adequately treated with adjuvant therapy and are currently disease free, and patients with stage I or II prostate cancer treated with prostatectomy or radiotherapy and are biochemically free of disease [for radical retropubic prostatectomy (RRP) prostate-specific antigen (PSA) < 0.3 and for radiotherapy PSA < 2.0 above the post treatment nadir])
* Any of the following:

  * Pregnant women
  * Women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, abstinence, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-07; Primary Completion 2011-06 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A. Pockaj, MD, Study Chair — Mayo Clinic Hospital
Locations (39):
- United States (39):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota

REFERENCES:
- [Result] Rule WG, Allred JB, Pockaj BA, Markovic SN, DiCaudo DJ, Erickson LA, Deming RL, Schild SE. Results of NCCTG N0275 (Alliance) - a phase II trial evaluating resection followed by adjuvant radiation therapy for patients with desmoplastic melanoma. Cancer Med. 2016 Aug;5(8):1890-6. doi: 10.1002/cam4.783. Epub 2016 Jul 1. PMID 27368067

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Adjuvant Radiation Therapy): Radiation therapy (RT) must begin within 8 weeks of surgical excision. Healing should be adequate to begin RT safely. Patients will receive a total of 30 Gy in 5 fractions of 6 Gy prescribed to Dmax, administered twice-a-week (Monday and Thursday or Tuesday and Friday) over approximately 2.5 weeks. Treatment will be administered with electrons only.
Period: Overall Study
Arm/Group | Treatment (Adjuvant Radiation Therapy)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Adjuvant Radiation Therapy)
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 68.0 [49.0 to 76.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: 2-year Local Recurrence Rate (LRR)/Incidence of Local Recurrence
Description: The primary endpoint is the incidence of local recurrence within 2 years after treatment. Local recurrence (LR) is defined as a desmoplastic melanoma lesion recurring within the radiated field. The properties of the binomial distribution will be used to construct a 95% confidence interval for the true 2-year local recurrence rate (LRR). The Kaplan-Meier method will be used if some patients are lost to follow-up.
Time Frame: Within 2 years after treatment
Measure: Number (95% Confidence Interval); unit: percentage of patients with LR
Arm/Group | Treatment (Adjuvant Radiation Therapy)
Number analyzed (Participants) | 20
percentage of patients with LR | 10 [0 to 23.2]

2. Secondary Outcome: Incidence of Regional and Systemic Metastases
Description: Incidence of regional and systemic metastasis: Incidences will be calculated for each cohort and 95% confidence intervals will be constructed using the properties of the binomial distribution.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Adjuvant Radiation Therapy)
Number analyzed (Participants) | 20
percentage of patients | 5 [0.1 to 24.9]

3. Secondary Outcome: Survival Time
Description: Survival time: Survival time is defined as the time from randomization to death due to any cause. The median survival time will be estimated using the method of Kaplan-Meier.
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval)
Arm/Group | Treatment (Adjuvant Radiation Therapy)
Number analyzed (Participants) | 20
Value | NA [NA to NA] — The median survival time was not reached.

4. Secondary Outcome: Failure Time
Description: Failure time is defined as the time from randomization to death due to any cause or disease progression. The median failure time will be estimated using the method of Kaplan-Meier.
Time Frame: Time from randomization to death due to any cause or disease progression (up to 5 years)
Measure: Median (95% Confidence Interval)
Arm/Group | Treatment (Adjuvant Radiation Therapy)
Number analyzed (Participants) | 20
Value | NA [NA to NA] — The median failure time was not reached.

5. Secondary Outcome: Toxicity
Description: For this secondary endpoint, toxicity is defined as a grade 3 or higher adverse events that is classified as either possibly, probably, or definitely related to study treatment. The assignment of attribution to study treatment and grade (or degree of severity) of the adverse event are classified using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 2.0. The number of participants reporting a grade 3 or higher toxicity are reported. For a list of all reported adverse events, please refer to the Adverse Events Section below.
Time Frame: Up to 5 years
Measure: Number; unit: number of participants
Arm/Group | Treatment (Adjuvant Radiation Therapy)
Number analyzed (Participants) | 20
number of participants | 0

6. Secondary Outcome: Change in Fatigue From Baseline to 3 Months as Assessed by the Brief Fatigue Inventory
Description: Fatigue Assessment: A portion of the Brief Fatigue Inventory will be used to determine fatigue changes throughout the course of radiation. Patients will fill out the questionnaire at baseline, weekly during radiation, and 3 months after the beginning of radiation. Fatigue will be defined as: minor if the patient answers 0-3 (on a 10 point scale), mild for answers of 4-6, and severe for answers of 7-10. The percentage of patients that have worsened (improved) fatigue from baseline to the radiation stage will be calculated. We will also compare fatigue levels at baseline to the 3 month visit. Worsened fatigue is defined as going from minor to mild, minor to severe, or mild to severe. Improved fatigue is defined as going from severe to mild, severe to minor, or mild to minor.
Time Frame: Baseline to up to 3 months
Measure: Number; unit: percentage of participants analyzed
Groups:
- Treatment (Adjuvant Radiation Therapy) Q01: Radiation therapy (RT) must begin within 8 weeks of surgical excision. Healing should be adequate to begin RT safely. Patients will receive a total of 30 Gy in 5 fractions of 6 Gy prescribed to Dmax, administered twice-a-week (Monday and Thursday or Tuesday and Friday) over approximately 2.5 weeks. Treatment will be administered with electrons only. Patients completed question 1 (Q01) of the Brief Fatigue Inventory (BFI) which instructs "Please rate your fatigue (weariness, tiredness) by circling the one number that best describes your fatigue right NOW."
- Treatment (Adjuvant Radiation Therapy) Q02: Radiation therapy (RT) must begin within 8 weeks of surgical excision. Healing should be adequate to begin RT safely. Patients will receive a total of 30 Gy in 5 fractions of 6 Gy prescribed to Dmax, administered twice-a-week (Monday and Thursday or Tuesday and Friday) over approximately 2.5 weeks. Treatment will be administered with electrons only. Patients completed question 2 (Q02) of the Brief Fatigue Inventory (BFI) which instructs "Please rate your fatigue (weariness, tiredness) by circling the one number that best describes your USUAL level of fatigue during the past 24 hours."
- Treatment (Adjuvant Radiation Therapy) Q03: Radiation therapy (RT) must begin within 8 weeks of surgical excision. Healing should be adequate to begin RT safely. Patients will receive a total of 30 Gy in 5 fractions of 6 Gy prescribed to Dmax, administered twice-a-week (Monday and Thursday or Tuesday and Friday) over approximately 2.5 weeks. Treatment will be administered with electrons only. Patients completed question 3 (Q03) of the Brief Fatigue Inventory (BFI) which instructs "Please rate your fatigue (weariness, tiredness) by circling the one number that best describes your WORST level of fatigue during the past 24 hours."
Arm/Group | Treatment (Adjuvant Radiation Therapy) Q01 | Treatment (Adjuvant Radiation Therapy) Q02 | Treatment (Adjuvant Radiation Therapy) Q03
Number analyzed (Participants) | 17 | 17 | 17
percentage of participants analyzed
  Improve | 11.8 | 23.5 | 29.4
  Same | 76.5 | 64.7 | 64.7
  Worsened | 11.8 | 11.8 | 5.9

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at the end of radiation therapy (RT) every 3 months for 3 years and then every 6 months for 2 more years; Up to 5 years.
Description: This study will utilize the Common Toxicity Criteria (CTC) version 2.0 for adverse event monitoring and reporting. All graded adverse events are reported.
Arm/Group | Treatment (Adjuvant Radiation Therapy)
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 18/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Adjuvant Radiation Therapy) (N=20)
Cardiac disorder (Cardiac disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Pain due to radiation (General disorders) | 5 (8)
Dermatitis radiation (Injury, poisoning and procedural complications) | 18 (28)
INR increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes